CLINICAL TRIAL: NCT00125008
Title: Randomized Controlled Evaluation of the Vi Polysaccharide Vaccine Against Typhoid Fever in Eastern Kolkata, West Bengal, India
Brief Title: Evaluation of the Vi Polysaccharide Vaccine Against Typhoid Fever
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: National Institute of Cholera and Enteric Diseases, India (Other); Wellcome Trust (Other); University of Western Ontario, Canada (Other); GlaxoSmithKline (Industry)
Responsible Party: Mr. Leon Ochiai, International Vaccine Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: T-17
Record Dates: First submitted 2005-07-28; First posted 2005-07-29 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Typhoid; Paratyphoid Fever
Keywords: Salmonella; Typhoid vaccine; enteric fever
MeSH Terms: conditions — Typhoid Fever; Paratyphoid Fever | interventions — Vi polysaccharide vaccine, typhoid; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Typhoid Vi vaccine
  Interventions: Biological: Typhoid Vi vaccine
- 2 (Active Comparator): Hepatitis A vaccine
  Interventions: Biological: Hepatitis A vaccine

INTERVENTIONS:
Biological: Typhoid Vi vaccine — single 0.5ml dose (25ug of purified Vi polysaccharide of S. typhi)
  Other Names: Typherix
  Arms: 1
Biological: Hepatitis A vaccine — 720 EL.U. of inactivated hepatitis A viral antigen for children 1440 EL.U. of inactivated hepatitis A viral antigen for adults
  Other Names: Havrix
  Arms: 2

SUMMARY:
This study is part of the International Vaccine Institute's (IVI's) typhoid Vi demonstration project that aims to accelerate the rational introduction of Vi vaccines in typhoid endemic countries. The purpose of this study is to determine the effectiveness of the Vi vaccine following a mass typhoid immunization campaign in an endemic area in Kolkata, India. The cost-effectiveness of the Vi vaccination and the logistic feasibility of a mass typhoid immunization campaign will also be evaluated.

DETAILED DESCRIPTION:
Typhoid fever is a major cause of morbidity worldwide. The disease predominantly affects school-aged children, is more prevalent in urban areas, may last for several weeks and can lead to serious complications. Management of this disease is further complicated by the emergence of multi-drug resistant strains. Vaccination of high risk populations is considered the most promising strategy for the control of typhoid fever. The Vi polysaccharide vaccine has been targeted for accelerated introduction into public health programs since it has been shown to have consistent efficacy results even in areas of high typhoid incidence, is given as a single dose, lacks patent protection and requires less strict cold chain requirements.

This project attempts to evaluate a new vaccination strategy for residents of endemic areas. A cluster-randomized trial involving the Vi polysaccharide vaccine and an active control (Hepatitis A) was designed to determine the effectiveness and the feasibility of providing Vi vaccine under actual programmatic conditions in 2 contiguous urban wards in Kolkata. The vaccines used in this study are internationally produced and locally licensed. A 1 year pilot phase will precede the actual Vi-demonstration project. Surveillance for typhoid fever cases will continue after the mass immunization campaign. A passive surveillance system to evaluate adverse events following immunization will be implemented. Socio-economic studies will be conducted in parallel to the effectiveness evaluation. The knowledge, attitudes, beliefs and practices among parents and health care providers regarding typhoid illness, treatment and prevention will be assessed. Logistic, feasibility and vaccine costs will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the project census
* Age >=2 years
* Provide informed consent to receive vaccine

Exclusion Criteria:

* Fever (>37.5 degrees Celsius)
* Pregnancy
* Lactating

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37673 (Actual)
Dates: Start 2003-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Total protection against S. typhi | 2 years from zero time

SECONDARY OUTCOMES:
Indirect protection against S. typhi | 2 years from zero time
Overall protection against S. typhi | 2 years from zero time
Total protection against S. paratyphi | 2 years from zero time
Adverse event(s) following immunization | 30 days from vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Sujit K Bhatttacharya, MD, Principal Investigator — National Institute of Cholera and Enteric Diseases, India
Locations (1):
- National Institute of Cholera and Enteric Diseases, Kolkata, West Bengal, India

REFERENCES:
- [Background] Acosta CJ, Galindo CM, Ochiai RL, Danovaro-Holliday MC, Page AL, Thiem VD, Park JK, Park E, Koo H, Wang XY, Abu-Elyazeed R, Ali M, Albert MJ, Ivanoff B, Pang T, Xu ZY, Clemens JD. The role of epidemiology in the introduction of vi polysaccharide typhoid fever vaccines in Asia. J Health Popul Nutr. 2004 Sep;22(3):240-5. PMID 15609776
- [Background] Dutta S, Sur D, Manna B, Bhattacharya SK, Deen JL, Clemens JD. Rollback of Salmonella enterica serotype Typhi resistance to chloramphenicol and other antimicrobials in Kolkata, India. Antimicrob Agents Chemother. 2005 Apr;49(4):1662-3. doi: 10.1128/AAC.49.4.1662-1663.2005. No abstract available. PMID 15793167
- [Derived] Sur D, Ochiai RL, Bhattacharya SK, Ganguly NK, Ali M, Manna B, Dutta S, Donner A, Kanungo S, Park JK, Puri MK, Kim DR, Dutta D, Bhaduri B, Acosta CJ, Clemens JD. A cluster-randomized effectiveness trial of Vi typhoid vaccine in India. N Engl J Med. 2009 Jul 23;361(4):335-44. doi: 10.1056/NEJMoa0807521. PMID 19625715